CLINICAL TRIAL: NCT01798030
Title: Association of Vitamin D With Diabetes, Osteoporosis and Cardiovascular Risk
Brief Title: Vitamin D Retrospective Study and Role With Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alice S. Ryan, PhD, Professor, Baltimore VA Medical Center
Other Study IDs: 43973
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Vitamin D Status; Glucose Tolerance; Blood Pressure; Bone Mineral Density; Hyperlipidemia
Keywords: Vitamin D; Diabetes; Osteoporosis; Cardiovascular Risk
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus; Osteoporosis | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Vitamin D, IGF-1, and PTH levels will be measured in coded plasma samples belonging to the PI and collaborating Investigators within the GRECC that are stored in our freezers (from previously approved studies: HP-00040261,HP-00040975, HP-00041166 and HP-00041199) . The Nutrition Obesity research center genetics core will determine Vitamin D receptor polymorphisms on de-identified samples. No clinical information will accompany the samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitamin D: Specimen analysis
  Interventions: Other: Vitamin D

INTERVENTIONS:
Other: Vitamin D — N/A, frozen specimen study

SUMMARY:
Vitamin D deficiency is associated with a heightened risk for developing type 2 diabetes, hypertension, and osteopenia/osteoporosis. Vitamin D is made in the skin when it is exposed to sunlight and it is also obtained from the diet and dietary supplements. Older people, individuals with high skin pigmentation, obese and sedentary individuals have low levels of Vitamin D because pigmentation blocks Vitamin D production in the skin, aging and physical inactivity are associated with reduced exposure to sunlight, and obesity is associated with the storage of Vitamin D in fat preventing its utilization by muscle, bone and other tissues that require its metabolic action. These conditions are also associated with heightened risk for developing type 2 diabetes, glucose intolerance, hypertension, and osteopenia/osteoporosis in older and obese individuals. This is particularly heightened in older women who tend to have increased body fat, are more physically inactive and are at high risk for central obesity and its metabolic consequences of diabetes, hypertension and osteoporosis.

DETAILED DESCRIPTION:
The heightened prevalence of obesity in aging especially in postmenopausal women suggests that interventions to raise Vitamin D levels might be preventive of these diseases. Investigators have completed studies of the effects of weight loss and exercise interventions in approximately 400 older women and men over the last 15 years, many of whom are obese. Investigators have data on glucose tolerance, blood pressure and bone density in these studies and stored plasma in which investigators can analyze Vitamin D levels. Vitamin D may be an important risk factor for these metabolic diseases and the availability of these samples for Vitamin D analysis will allow investigators to perform a cross-sectional study to address relationships of Vitamin D levels to glucose intolerance and diabetes, hypertension/blood pressure status, bone mineral density, the degree of obesity, and physical activity status measured as maximal aerobic capacity and accelerometry in these older men and women.

The results of this study have the potential to impact clinical practice in the prevention and treatment of diabetes, hypertension, and osteopenia/osteoporosis. This would circumvent the current dilemma for prevention of these chronic diseases through treatment of obesity, as these data would provide immediate prospects for changing the recommended doses of Vitamin D beneficial for reducing risk for these diseases.

The purpose of this study is to 1) determine the prevalence of Vitamin D deficiency in obese, older men and postmenopausal women and 2) the association of Vitamin D levels to glucose tolerance, blood pressure, bone mineral density, and hyperlipidemia, as well as association with Vitamin D receptor gene polymorphisms affecting metabolic responses to Vitamin D.

ELIGIBILITY:
Inclusion Criteria: 45-85 years of age

Exclusion Criteria: none

-

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese, older men and postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2009-11; Primary Completion 2021-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Vitamin D | Day 1
  Vitamin D level ng/dl

OTHER OUTCOMES:
IGF-1 | Day 1
  Insulin like growth factor
IGF binding proteins | Day 1
  Insulin Growth Factor Binding protein levels
PTH | Day 1
  Parathyroid Hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Ryan, PhD, Principal Investigator — Baltimore VAMC
Locations (1):
- Baltimore VAMC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorkin JD, Vasaitis TS, Streeten E, Ryan AS, Goldberg AP. Evidence for threshold effects of 25-hydroxyvitamin D on glucose tolerance and insulin resistance in black and white obese postmenopausal women. J Nutr. 2014 May;144(5):734-42. doi: 10.3945/jn.114.190660. Epub 2014 Apr 9. PMID 24717362